## atlas: An Interactive Text Messaging Program Combining Weather Alerts With Hyper-Localized Resources & Actionable Insights for Addressing Climate Change NCT06995755

Unique Protocol ID: R43ES035344 November 6, 2024

## INFORMED CONSENT FORM

Title of Research: atlas

**Principal Investigator**: Sara Johnson, Ph.D.

**Address**: ProChange Behavior Solutions 91 Point Judith Road, STE 26, Unit 333

Narragansett, RI 02882

Telephone: (888) 280-2516

## DESCRIPTION OF THE RESEARCH AND THE RIGHTS OF PARTICIPANTS

## **Key Information:**

- The purpose of the study is to test *atlas*, a new text messaging program designed to give people information about extreme weather events and climate change.
- If you choose to participate, you will be asked to use *atlas* for 30 days and to complete a survey at the end to tell us what you thought about it.
- Risks or discomforts from this research include possible discomfort answering some questions and the time you spend using the program. Your phone carrier may charge standard message and data rates for the text messages.
- The study will have no direct benefit to you. The results of this study may help us improve the program so it can help other people take steps to protect themselves from extreme weather events and to reduce climate change.
- You will be given a \$35 gift card as a thank you for joining the program and a \$40 gift card as a thank you for your time after you complete the survey 30 days later.
- You will be provided a copy of this consent form.
- Taking part in this research project is voluntary. You don't have to take part and you can stop it at any time.

If you have any questions, you can call (888) 280-2516. Dr. Sara Johnson, the person who is leading this study, will discuss them with you. ProChange Behavior Solutions is a company that designs programs to help people make positive changes in their lives. It is located in Rhode Island.

- 1) <u>Purpose of Study</u>: The purpose of this research is to get feedback on a new text messaging program to give people information about extreme weather events and climate change. Your input will help us develop a text messaging program that people find helpful and easy to use.
  - What You Are Being Asked to Do: You are one of 50 individuals in Rhode Island who are being asked to take part in this research. You do not have to go anywhere to take part in the study. You can text the phone number we provide to see if you are eligible. If you are invited to use atlas, you will have access to the text messaging program for 30 days. Thirty days after you sign up, we will invite you to

complete a survey to tell us what you think about *atlas*. The time people spend using *atlas* will vary, but most people will spend less than a total of 2 hours using the program over the 30 days.

You will receive a \$35 gift card after you finish the first session of *atlas* and a \$40 gift card after you complete the survey 30 days later.

- 2) <u>Risks</u>: You may find that some of the questions make you uneasy and that you don't want to answer them. That's OK. You can stop answering questions at any time. If you want to talk to someone about questions or concerns later, please reach out to the Rhode Island State Climate Office at 401-222-1360 ext. 77041, the Rhode Island Department of Environmental Management at <u>401-222-4700</u>, ext. 2772409, or a person you trust.
- **Benefits**: The information gathered in this research will help us improve the *atlas* text messaging program to help people take steps to protect themselves in extreme weather and to reduce climate change. Some people may find that taking part in this project is interesting and helpful.
- 4) <u>Costs/Payment</u>: There is no cost to you. This project is funded by the National Institute of Environmental Health Sciences. Costs of all services and materials will be covered by a grant awarded to Pro-Change Behavior Solutions, Inc. You will receive a \$35 gift card after you finish the first session of *atlas* and a \$40 gift card when you take the 30-day survey.
- 5) <u>Confidentiality</u>: The Information you provide to atlas will be kept private and used only for research purposes. Your name will not be associated with your answers to the text messaging program. There is one exception to the promise of confidentiality. If we see or are told that someone is being abused or neglected or that someone is planning to harm themselves or someone else, we will disclose this information to the proper authorities.
- **Right to Refuse to Participate**: You have the right to refuse to take part in this research, and to stop taking part at any time. Your choice about taking part in this research will in no way impact your relationship with ProChange.

**Questions/Concerns**: This research study is being conducted by Pro-Change Behavior Solutions. If you have any questions or concerns about this research, please contact the study lead, Sara Johnson, at sjohnson@prochange.com, or call (401) 360-2980.

If you have questions or concerns about your rights as a research participant, if this study causes you any harm, or if you feel you are receiving pressure to continue in this research against your wishes, please call the ProChange Institutional Review Board Chairperson, Dr. Ted Myatt, at (401) 489-8332.

I have read the consent form and have no further questions about taking part in this project at this time. I understand that I may ask any other questions later, that taking part is voluntary, and that I may withdraw from this project at any time. By texting back yes, I agree to take part in this research study.